CLINICAL TRIAL: NCT01881373
Title: Children's Healthy Living Program for Remote Underserved Minority Populations in the Pacific Region
Brief Title: Children's Healthy Living Community Randomized Trial
Acronym: CHL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: University of Guam (Other); Northern Marianas College (Unknown); University of Alaska Fairbanks (Other); American Samoa Community College (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: USDA 2011-68001-30335; 2011-68001-30335 (Other Grant/Funding Number: USDA/NIFA/AFRI); 2018-69001-27551 (Other Grant/Funding Number: USDA/NIFA/AFRI)
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Results first posted 2020-05-01 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2023-06

CONDITIONS: Obesity; Acanthosis Nigricans; Central Obesity
Keywords: Obesity; Child; Food; Physical Activity; Pacific
MeSH Terms: conditions — Obesity; Acanthosis Nigricans; Obesity, Abdominal; Motor Activity

STUDY DESIGN:
Intervention Model Description: Community randomized intervention for child obesity prevention with multiple levels and components (policy, environment, messaging, and capacity)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CHL program (Experimental): Multiple component environmentally focused intervention designed with a community engagement process.
  Interventions: Other: CHL program
- Delayed Optimized CHL program (Other): Comparison community that participated in community engagement process and received delayed optimized program.
  Interventions: Other: Delayed Optimized CHL program
- Temporal (No Intervention): Communities assessed for temporal trends in anthropometry.

INTERVENTIONS:
Other: CHL program — Multiple component environmentally focused program designed with community engagement.
  Arms: CHL program
Other: Delayed Optimized CHL program — CHL programs with fewer component and shorter duration.
  Arms: Delayed Optimized CHL program

SUMMARY:
The goal is to build social/cultural, political/economic, and physical/built environments that will promote active play and intake of healthy food to prevent young child obesity in the Pacific Region. Our methods will support local culture in order to achieve this goal in these remote, underserved native populations. CHL will engage the community, and focus on capacity building and sustainable environmental change.

The focus of the CHL community-based program is to promote healthy eating and to increase physical activity. In order to demonstrate effectiveness, the investigators will recruit and measure children in six communities selected in each of our jurisdictions in the Pacific. These represent intervention communities, comparison communities, and temporal communities.

DETAILED DESCRIPTION:
The specific objectives of our study are as follows.

Objective. Decrease the prevalence of young child overweight and obesity; and its functional outcomes (decrease acanthosis nigricans, and increase sleep; increase moderate to vigorous physical activity and decrease sedentary behavior (screen time); increase healthy eating (fruit and vegetable intake, water intake; decrease sweetened beverage intake), through community-based primary prevention environmental interventions in the Pacific region.

Objective. Measure 2-8-year-old children at baseline and 24 months in selected communities to track behaviors and anthropometry that indicate healthy eating, physical activity, and BMI.

Objective. Measure 2-8 year old children at 78 months in the selected communities to determine the long term effect of the CHL program.

ELIGIBILITY:
Inclusion Criteria:

* Community criteria

Four (4) to six (6) communities in each of five (5) jurisdictions (Alaska, American Samoa, Commonwealth of Northern Mariana Islands, Guam & Hawai'i) chosen for community randomized program based on:

* 2000 U.S. Census criteria

  * >1000 people
  * >25% Native population,
  * >10% under 5y
* CHL Staff Community Evaluation

  * Sufficient Head Start/preschool, kindergarten
  * Children live & go to school in area
  * Separation between communities to allow testing
  * Access for CHL
  * Sufficient community cohesiveness
  * Sufficient settings for program (community centers, parks, stores…)
* Child criteria • 2-10 years of age

Exclusion Criteria:

* Child criteria

  * Known orthopedic, psychological or neurologic impairments that prevent physical activity
  * Presence or history of any metabolic or chronic health problems known to affect intermediary metabolism (e.g. untreated thyroid disease, cancer, hepatic disease, renal disease, diabetes, cardiovascular disease, hypertension)
  * Irregular use of prescription or over-the-counter medications known to affect appetite, food intake or intermediary metabolism (e.g. appetite suppressants, lithium, antidepressants, etc.)

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 9840 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Novotny, PhD, Principal Investigator — University of Hawaii
Locations (1):
- University of Hawaii, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: Yes
Request system whereby researchers submit a proposal, if approved by CHL steering committee, data is released using secure systems
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2017 to current
Access Criteria: citi training, approval of proposal by CHL program steering committee
URL: http://www.chl-pacific.org

REFERENCES:
- [Background] Fialkowski MK, DeBaryshe B, Bersamin A, Nigg C, Leon Guerrero R, Rojas G, Areta AA, Vargo A, Belyeu-Camacho T, Castro R, Luick B, Novotny R; CHL Team. A community engagement process identifies environmental priorities to prevent early childhood obesity: the Children's Healthy Living (CHL) program for remote underserved populations in the US Affiliated Pacific Islands, Hawaii and Alaska. Matern Child Health J. 2014 Dec;18(10):2261-74. doi: 10.1007/s10995-013-1353-3. PMID 24043557
- [Background] Wilken LR, Novotny R, Fialkowski MK, Boushey CJ, Nigg C, Paulino Y, Leon Guerrero R, Bersamin A, Vargo D, Kim J, Deenik J. Children's Healthy Living (CHL) Program for remote underserved minority populations in the Pacific region: rationale and design of a community randomized trial to prevent early childhood obesity. BMC Public Health. 2013 Oct 9;13:944. doi: 10.1186/1471-2458-13-944. PMID 24107083
- [Background] Novotny R, Fialkowski MK, Areta AA, Bersamin A, Braun K, DeBaryshe B, Deenik J, Dunn M, Hollyer J, Kim J, Leon Guerrero RT, Nigg CR, Takahashi R, Wilkens LR. University of Hawai'i Cancer Center Connection: The Pacific Way to Child Wellness: The Children's Healthy Living Program for Remote Underserved Minority Populations of the Pacific Region (CHL). Hawaii J Med Public Health. 2013 Nov;72(11):406-8. No abstract available. PMID 24251089
- [Background] Braun KL, Nigg CR, Fialkowski MK, Butel J, Hollyer JR, Barber LR, Bersamin A, Coleman P, Teo-Martin U, Vargo AM, Novotny R. Using the ANGELO model to develop the children's healthy living program multilevel intervention to promote obesity preventing behaviors for young children in the U.S.-affiliated Pacific Region. Child Obes. 2014 Dec;10(6):474-81. doi: 10.1089/chi.2014.0102. PMID 25369548
- [Background] Novotny R, Fialkowski MK, Li F, Paulino Y, Vargo D, Jim R, Coleman P, Bersamin A, Nigg CR, Leon Guerrero RT, Deenik J, Kim JH, Wilkens LR. Systematic Review of Prevalence of Young Child Overweight and Obesity in the United States-Affiliated Pacific Region Compared With the 48 Contiguous States: The Children's Healthy Living Program. Am J Public Health. 2015 Jan;105(1):e22-e35. doi: 10.2105/AJPH.2014.302283. PMID 25393168
- [Background] Fialkowski MK, Delormier T, Hattori-Uchima M, Leslie JH, Greenberg J, Kim JH, Deenik JL, Dunn MA, Areta IA, Novotny R. Children's Healthy Living Program (CHL) Indigenous Workforce Training to Prevent Childhood Obesity in the Underserved U.S. Affiliated Pacific Region. J Health Care Poor Underserved. 2015 May;26(2 Suppl):83-95. doi: 10.1353/hpu.2015.0054. PMID 25981090
- [Background] Butel J, Braun KL, Novotny R, Acosta M, Castro R, Fleming T, Powers J, Nigg CR. Assessing intervention fidelity in a multi-level, multi-component, multi-site program: the Children's Healthy Living (CHL) program. Transl Behav Med. 2015 Dec;5(4):460-9. doi: 10.1007/s13142-015-0334-z. Epub 2015 Aug 4. PMID 26622918
- [Background] Li F, Wilkens LR, Novotny R, Fialkowski MK, Paulino YC, Nelson R, Bersamin A, Martin U, Deenik J, Boushey CJ. Anthropometric measurement standardization in the US-affiliated pacific: Report from the Children's Healthy Living Program. Am J Hum Biol. 2016 May;28(3):364-71. doi: 10.1002/ajhb.22796. Epub 2015 Oct 12. PMID 26457888
- [Background] Aflague TF, Leon Guerrero RT, Delormier T, Novotny R, Wilkens LR, Boushey CJ. Examining the Influence of Cultural Immersion on Willingness to Try Fruits and Vegetables among Children in Guam: The Traditions Pilot Study. Nutrients. 2019 Dec 20;12(1):18. doi: 10.3390/nu12010018. PMID 31861756
- [Background] Yamanaka AB, Davis JD, Wilkens LR, Hurwitz EL, Fialkowski MK, Deenik J, Leon Guerrero RT, Novotny R. Determination of Child Waist Circumference Cut Points for Metabolic Risk Based on Acanthosis Nigricans, the Children's Healthy Living Program. Prev Chronic Dis. 2021 Jun 24;18:E64. doi: 10.5888/pcd18.210021. PMID 34166179
- [Background] Butel J, Braun KL. The Role of Collective Efficacy in Reducing Health Disparities: A Systematic Review. Fam Community Health. 2019 Jan/Mar;42(1):8-19. doi: 10.1097/FCH.0000000000000206. PMID 30431465
- [Background] Leon Guerrero RT, Barber LR, Aflague TF, Paulino YC, Hattori-Uchima MP, Acosta M, Wilkens LR, Novotny R. Prevalence and Predictors of Overweight and Obesity among Young Children in the Children's Healthy Living Study on Guam. Nutrients. 2020 Aug 20;12(9):2527. doi: 10.3390/nu12092527. PMID 32825433
- [Background] Novotny R, Earle ME, Jung YO, Julian GJ, Hill E, Leon Guerrero RT, Coleman P, Deenik J, Boushey C, Wilkens LR. University of Hawai'i Cancer Center Connection: Pacific Tracker (PacTrac) Version 3.1 Diet and Physical Activity Assessment Tool for the Pacific Region. Hawaii J Health Soc Welf. 2021 Jul;80(7):165-168. PMID 34278324
- [Background] Greenberg JA, Luick B, Alfred JM, Barber LR Jr, Bersamin A, Coleman P, Esquivel M, Fleming T, Leon Guerrero RT, Hollyer J, Johnson EL, Novotny R, deBlair Remengesau S, Yamanaka A. The Affordability of a Thrifty Food Plan-based Market Basket in the United States-affiliated Pacific Region. Hawaii J Health Soc Welf. 2020 Jul 1;79(7):217-223. PMID 32666055
- [Background] Yonemori KM, Ennis T, Novotny R, Fialkowski MK, Ettienne R, Wilkens LR, Leon Guerrero RT, Bersamin A, Coleman P, Li F, Boushey CJ. Collecting wrappers, labels, and packages to enhance accuracy of food records among children 2-8 years in the Pacific region: Children's Healthy Living Program (CHL). J Food Compost Anal. 2017 Dec;64(Pt 1):112-118. doi: 10.1016/j.jfca.2017.04.012. Epub 2017 Apr 23. PMID 29398780
- [Background] Paulino YC, Ettienne R, Novotny R, Wilkens LR, Shomour M, Sigrah C, Remengesau SD, Johnson EL, Alfred JM, Gilmatam DF. Areca (betel) nut chewing practices of adults and health behaviors of their children in the Freely Associated States, Micronesia: Findings from the Children's Healthy Living (CHL) Program. Cancer Epidemiol. 2017 Oct;50(Pt B):234-240. doi: 10.1016/j.canep.2017.07.009. PMID 29120830
- [Background] Novotny R, Li F, Leon Guerrero R, Coleman P, Tufa AJ, Bersamin A, Deenik J, Wilkens LR. Dual burden of malnutrition in US Affiliated Pacific jurisdictions in the Children's Healthy Living Program. BMC Public Health. 2017 May 22;17(1):483. doi: 10.1186/s12889-017-4377-6. PMID 28532446
- [Background] Yamanaka A, Fialkowski MK, Wilkens L, Li F, Ettienne R, Fleming T, Power J, Deenik J, Coleman P, Leon Guerrero R, Novotny R. Quality assurance of data collection in the multi-site community randomized trial and prevalence survey of the children's healthy living program. BMC Res Notes. 2016 Sep 2;9(1):432. doi: 10.1186/s13104-016-2212-2. PMID 27590179
- [Background] Novotny R, Li F, Fialkowski MK, Bersamin A, Tufa A, Deenik J, Coleman P, Guerrero RL, Wilkens LR; Children's Healthy Living (CHL) Program. Prevalence of obesity and acanthosis nigricans among young children in the children's healthy living program in the United States Affiliated Pacific. Medicine (Baltimore). 2016 Sep;95(37):e4711. doi: 10.1097/MD.0000000000004711. PMID 27631218
- [Background] Fialkowski MK, Yamanaka A, Wilkens LR, Braun KL, Butel J, Ettienne R, McGlone K, Remengesau S, Power JM, Johnson E, Gilmatam D, Fleming T, Acosta M, Belyeu-Camacho T, Shomour M, Sigrah C, Nigg C, Novotny R. Recruitment Strategies and Lessons Learned from the Children's Healthy Living Program Prevalence Survey. AIMS Public Health. 2016 Mar 21;3(1):140-157. doi: 10.3934/publichealth.2016.1.140. eCollection 2016. PMID 29546153
- [Background] Esquivel MK, Nigg CR, Fialkowski MK, Braun KL, Li F, Novotny R. Influence of Teachers' Personal Health Behaviors on Operationalizing Obesity Prevention Policy in Head Start Preschools: A Project of the Children's Healthy Living Program (CHL). J Nutr Educ Behav. 2016 May;48(5):318-325.e1. doi: 10.1016/j.jneb.2016.02.007. PMID 27169640
- [Background] Esquivel M, Nigg CR, Fialkowski MK, Braun KL, Li F, Novotny R. Head Start Wellness Policy Intervention in Hawaii: A Project of the Children's Healthy Living Program. Child Obes. 2016 Feb;12(1):26-32. doi: 10.1089/chi.2015.0071. Epub 2016 Jan 15. PMID 26771119
- [Result] Novotny R, Davis J, Butel J, Boushey CJ, Fialkowski MK, Nigg CR, Braun KL, Leon Guerrero RT, Coleman P, Bersamin A, Areta AAR, Barber LR Jr, Belyeu-Camacho T, Greenberg J, Fleming T, Dela Cruz-Talbert E, Yamanaka A, Wilkens LR. Effect of the Children's Healthy Living Program on Young Child Overweight, Obesity, and Acanthosis Nigricans in the US-Affiliated Pacific Region: A Randomized Clinical Trial. JAMA Netw Open. 2018 Oct 5;1(6):e183896. doi: 10.1001/jamanetworkopen.2018.3896. PMID 30646266
- [Result] Butel J, Braun KL, Nigg CR, Leon Guerrero R, Fleming T, Bersamin A, Coleman P, Novotny R. Estimating intervention dose of the multilevel multisite children's healthy living program intervention. Transl Behav Med. 2020 Oct 8;10(4):989-997. doi: 10.1093/tbm/ibz073. PMID 31116404
- [Result] Gittelsohn J, Novotny R, Trude ACB, Butel J, Mikkelsen BE. Challenges and Lessons Learned from Multi-Level Multi-Component Interventions to Prevent and Reduce Childhood Obesity. Int J Environ Res Public Health. 2018 Dec 24;16(1):30. doi: 10.3390/ijerph16010030. PMID 30586845
- [Result] Korn AR, Butel J, Davis J, Yamanaka AB, Coleman P, Wilkens LR, Economos CD, Novotny R. Role of social ecological model level on young Pacific children's sugar-sweetened beverage and water intakes: Children's Healthy Living intervention. Public Health Nutr. 2021 Jun;24(8):2318-2323. doi: 10.1017/S1368980020004796. Epub 2020 Nov 25. PMID 33234187
- [Derived] Dumuid D, Yamanaka AB, Chong KH, Okely AD, Wilkens LR, Shvetsov YB, Lozano CP, Novotny R. Diet, Activity and Sleep Clusters Associated With Obesity Markers of Children in the US-Affiliated Pacific. Acta Paediatr. 2025 Jul;114(7):1642-1652. doi: 10.1111/apa.70012. Epub 2025 Feb 24. PMID 39989394
- [Derived] Novotny R, Yamanaka AB, Butel J, Boushey CJ, Dela Cruz R, Aflague T, Coleman P, Shallcross L, Fleming T, Wilkens LR. Maintenance Outcomes of the Children's Healthy Living Program on Overweight, Obesity, and Acanthosis Nigricans Among Young Children in the US-Affiliated Pacific Region: A Randomized Clinical Trial. JAMA Netw Open. 2022 Jun 1;5(6):e2214802. doi: 10.1001/jamanetworkopen.2022.14802. PMID 35666503
- See also: CHL program website — http://www.chl-pacific.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: communities were selected where >25% of the population was of indigenous/native descent (native to each jurisdiction), >10% of the population was under age 10 years, >1000 population size, and communities were relatively accessible
Pre-assignment Details: Eighteen selected communities were matched for size and randomized within jurisdiction to intervention or control. Nine additional communities were monitored with no randomization for temporal trends of obesity. 2-8 year old children and their households and environments were measured and evaluated in each of these communities.
Units Other Than Participants: Communities
Groups:
- Temporal: Communities assessed for temporal trends
Period: Baseline
Arm/Group | CHL Program | Delayed Optimized CHL Program | Temporal
Started (community randomized trial with 2 cross sectional samples at baseline and 24 months.) | 1517; 9 Communities (The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.) | 1491; 9 Communities (The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.) | 1321; 9 Communities (The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.)
Completed | 1517; 9 Communities (The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.) | 1491; 9 Communities (The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.) | 1321; 9 Communities (The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.)
Not Completed | 0; 0 Communities | 0; 0 Communities | 0; 0 Communities
Period: 24 Months
Arm/Group | CHL Program | Delayed Optimized CHL Program | Temporal
Started | 1342; 9 Communities (The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.) | 1295; 9 Communities (The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.) | 1405; 9 Communities (The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.)
Completed | 1342; 9 Communities (The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.) | 1295; 9 Communities (The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.) | 1405; 9 Communities (The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.)
Not Completed | 0; 0 Communities | 0; 0 Communities | 0; 0 Communities
Period: 78 Months
Arm/Group | CHL Program | Delayed Optimized CHL Program | Temporal
Started | 500; 9 Communities (The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.) | 479; 9 Communities (The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.) | 490; 9 Communities (The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.)
Completed | 500; 9 Communities (The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.) | 479; 9 Communities (The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.) | 490; 9 Communities (The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.)
Not Completed | 0; 0 Communities | 0; 0 Communities | 0; 0 Communities

BASELINE CHARACTERISTICS:
Population: 2 to 8 year old children
Units Other Than Participants: community
Groups:
- Control Community: Control community that participated in community engagement process and received delayed optimized program.
- Temporal: Control community with limited interaction; for temporal change assessment of anthropometry.
- Total: Total of all reporting groups
Arm/Group | CHL Program | Control Community | Temporal | Total
Number analyzed (Participants) | 3359 | 3265 | 3216 | 9840
Number analyzed (community) | 9 | 9 | 9 | 27
Age, Continuous [Mean (Full Range); unit: years] | 5.42 [2 to 8] | 5.49 [2 to 8] | 5.22 [2 to 8] | 5.38 [2 to 8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1699 | 1596 | 1571 | 4866
  Male | 1660 | 1669 | 1645 | 4974
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 35 | 28 | 215 | 278
  Asian | 186 | 410 | 468 | 1064
  Native Hawaiian or Other Pacific Islander | 1940 | 1735 | 1281 | 4956
  Black or African American | 32 | 8 | 17 | 57
  White | 302 | 328 | 363 | 993
  More than one race | 842 | 735 | 848 | 2425
  Unknown or Not Reported | 22 | 21 | 24 | 67
Region of Enrollment [Count of Participants; unit: Participants] — Participants were from communities in 5 jurisdictions which were Commonwealth of the Northern Mariana Islands, Guam, American Samoa, Alaska and Hawaii. In this table, the United States represents Alaska and United States Minor Outlying Islands represents Hawaii.
  Participants
    Northern Mariana Islands | 714 | 688 | 717 | 2119
    Guam | 781 | 759 | 277 | 1817
    American Samoa | 682 | 673 | 739 | 2094
    United States | 433 | 425 | 736 | 1594
    United States Minor Outlying Islands | 749 | 720 | 747 | 2216

OUTCOME MEASURES:

1. Primary Outcome: Change in Prevalence of Overweight and Obesity Using Body Mass Index Percentile for Age and Sex
Description: Body mass index is weight in kg divided by height in meters squared. Overweight is > = 85th percentile to < 95th percentile BMI for age and sex according to CDC 2000. Obesity is > = 95th percentile BMI for age and sex according to CDC 2000. Change from baseline to 24 months in prevalence of overweight plus obesity in selected communities. Comparison group is healthy weight >= 5th percentile to < 85th percentile for age and sex according to CDC 2000. Underweight (<5th percentile) were excluded.
Time Frame: Baseline, 24 months
Population: Children 2-8y in selected communities of the Pacific Region; the children from each community recruited each time were NOT the same children. The number of communities is consistent across time.
Measure: Mean (Standard Error); unit: percentage of 2 to 8 yo children
Units Other Than Participants: communities
Groups:
- Control Community: Comparison community that participated in community engagement process and will receive delayed optimized program.
- Temporal: Communities measured for temporal trends
Arm/Group | CHL Program | Control Community | Temporal
Number analyzed (Participants) | 2859 | 2786 | 2726
Number analyzed (communities) | 9 | 9 | 9
percentage of 2 to 8 yo children | -2.8 (1.16) | 1.4 (1.49) | -0.40 (2.0)
Statistical Analysis 1: Comparison: CHL Program vs Control Community; Test type: Superiority — Hierarchical logistic model accounting for randomization of communities and clustering of children within communities in strata of jurisdictions weighted for number of children less than age 10 in communities. Chi-square test accounts for degrees of freedom based on number of communities; p = 0.02, Regression, Logistic; Hierarchical model; Mean Difference (Final Values) = -3.88, 95% CI 2-sided [-7.29 to -0.47] — Intervention vs control communities comparing 24 months to baseline
Statistical Analysis 2: Comparison: CHL Program vs Temporal; The children from each community recruited each time were NOT the same children. The number of communities is consistent across time; Test type: Superiority — The children from each community recruited each time were NOT the same children. The number of communities is consistent across time; p = 0.28, Regression, Logistic — The children from each community recruited each time were NOT the same children. The number of communities is consistent across time; The children from each community recruited each time were NOT the same children. The number of communities is consistent across time; Mean Difference (Final Values) = -2.63, 95% CI 2-sided [-8.58 to 3.32]

2. Primary Outcome: Change in Waist Circumference
Description: Waist circumference measured in centimeters at umbilicus.
Time Frame: Baseline, 78 months
Population: Children 2-8 years in the selected Pacific communities.The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.
Measure: Mean (Standard Error); unit: centimeters
Units Other Than Participants: communities
Arm/Group | CHL Program | Control Community | Temporal
Number analyzed (Participants) | 2017 | 1970 | 1811
Number analyzed (communities) | 9 | 9 | 9
centimeters | 0.83 (0.05) | 2.47 (0.04) | 1.19 (0.03)
Statistical Analysis 1: Comparison: CHL Program vs Control Community; [analysis description as in outcome 1, analysis 2]; Test type: Superiority — Hierarchical model accounting for randomization of communities and clustering of children within communities in strata of jurisdictions weighted for number of children less than age 10 in communities. Chi-square test accounts for degrees of freedom based on number of communities; p = 0.009, Regression, Linear — Intervention vs control communities comparing 78 months to baseline; Hierarchical model; Mean Difference (Final Values) = -1.64, 95% CI 2-sided [-2.87 to -0.41]
Statistical Analysis 2: Comparison: CHL Program vs Temporal; Intervention vs temporal comparing 78 months to baseline; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.49, Regression, Linear; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = 4.35, 95% CI 2-sided [-8.5 to 17.24]

3. Primary Outcome: Prevalence of Acanthosis Nigricans
Description: Scale title: Burke Acanthosis nigricans Score, minimum 0, maximum 4. Higher score is worse. Analysis was dichotomized as present (1-4) or absent (0).
  A Screening on back of neck for Acanthosis nigricans according to Burke, J., D. Hale, H. Hazuda, and M. Stern. 1999. A quantitative scale of acanthosis nigricans. Diabetes Care. 22(10):1655-1659. Epub 1999/10/20. PubMed PMID: 10526730. Scale varies from 0 to 4 with 0 as not present and 4 most severe. Analysis was done on absent (0) or present (1-4).
Time Frame: Baseline, 24 months
Population: Children 2-8 in communities that were randomized to intervention or control. Acanthosis nigricans not assessed in temporal communities.The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.
Measure: Mean (Standard Error); unit: percentage of 2-8 yo children
Units Other Than Participants: communities
Groups:
- Temporal Community: Community assessed for temporal change in anthropometry.
Arm/Group | CHL Program | Control Community | Temporal Community
Number analyzed (Participants) | 2859 | 2786 | 0
Number analyzed (communities) | 9 | 9 | 0
percentage of 2-8 yo children | -4.1 (0.79) | -0.5 (0.96) |
Statistical Analysis 1: Comparison: CHL Program vs Control Community; Intervention vs control comparing 24 months to baseline; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.01, Regression, Logistic; Hierarchical model; Difference in prevalence = -3.6

4. Primary Outcome: Change in Prevalence of Overweight and Obesity Using Body Mass Index Percentile for Age and Sex
Description: Body mass index is weight in kg divided by height in meters squared. Overweight is > = 85th percentile to < 95th percentile BMI for age and sex according to CDC 2000. Obesity is > = 95th percentile BMI for age and sex according to CDC 2000. Change from baseline to 78 months in prevalence of overweight plus obesity in selected communities. Comparison group is healthy weight >= 5th percentile to < 85th percentile for age and sex according to CDC 2000. Underweight (<5th percentile) were excluded.
Time Frame: Baseline, 78 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of 2 to 8 yo children
Units Other Than Participants: communities
Arm/Group | CHL Program | Control Community | Temporal
Number analyzed (Participants) | 2017 | 1970 | 1811
Number analyzed (communities) | 9 | 9 | 9
percentage of 2 to 8 yo children | -5.28 (0.17) | 7.32 (0.11) | -0.19 (0.11)
Statistical Analysis 1: Comparison: CHL Program vs Control Community; Intervention vs. control. The children from each community recruited each time were NOT the same children. The number of communities is consistent across time; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.003, Regression, Logistic — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 2]; change in prevalence between communities = -12.6, 95% CI 2-sided [-20.92 to -4.28] — The children from each community recruited each time were NOT the same children. The number of communities is consistent across time
Statistical Analysis 2: Comparison: CHL Program vs Temporal; Intervention vs. Temporal communities. The children from each community recruited each time were NOT the same children. The number of communities is consistent across time; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.33, Regression, Logistic — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -3.43, 95% CI 2-sided [-10.36 to 3.50]

5. Primary Outcome: Change in Waist Circumference
Description: Waist circumference measured in centimeters at umbilicus.
Time Frame: Baseline, 24 months
Population: Children 2-8 years in the selected Pacific communities. The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.
Measure: Mean (95% Confidence Interval); unit: centimeters
Units Other Than Participants: communities
Arm/Group | CHL Program | Control Community | Temporal
Number analyzed (Participants) | 2859 | 2786 | 2726
Number analyzed (communities) | 9 | 9 | 9
centimeters | -0.12 [-0.72 to 0.49] | 0.59 [0.33 to 0.85] | 0.54 [-0.14 to 1.21]
Statistical Analysis 1: Comparison: CHL Program vs Control Community; [analysis description as in outcome 1, analysis 2]; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.02, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-1.37 to -0.05] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: CHL Program vs Temporal; [analysis description as in outcome 1, analysis 2]; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.13, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.65, 95% CI 2-sided [-1.79 to 0.49]

6. Secondary Outcome: Change in Sugar Sweetened Beverage Intake
Description: cups per day, determined from 2 random days of food records and weighted for weekend and weekday
Time Frame: Change from baseline to 24 months
Population: Children 2 to 8 from communities randomized to CHL program or Control. Temporal communities not assessed for sugar sweetened beverage intake.The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.
Measure: Mean (Standard Error); unit: cups per day
Units Other Than Participants: communities
Arm/Group | CHL Program | Control Community | Temporal Community
Number analyzed (Participants) | 2859 | 2786 | 0
Number analyzed (communities) | 9 | 9 | 0
cups per day | -0.05 (0.08) | -0.06 (0.04) |
Statistical Analysis 1: Comparison: CHL Program vs Control Community; Intervention vs control comparing 24 months to baseline; Test type: Superiority — Hierarchical linear model accounting for randomization of communities and clustering of children within communities in strata of jurisdictions weighted for number of children less than age 10 in communities. Chi-square test accounts for degrees of freedom based on number of communities.The children from each community recruited each time were NOT the same children. The number of communities is consistent across time; p = 0.86, Regression, Linear; Hierarchical model; Mean Difference (Final Values) = 0.01

7. Secondary Outcome: Change in Mean of Moderate and Vigorous Activity Per Day in Minutes
Description: number of minutes per day within bouts of 5 minutes averaged over 4 to 6 days of accelerometer usage
Time Frame: Baseline, 24 months
Population: Children 2 to 8 randomized to CHL program or Control Community. Temporal community not assessed for physical activity.
Measure: Mean (Standard Error); unit: number of minutes per day within bouts o
Units Other Than Participants: communities
Arm/Group | CHL Program | Control Community | Temporal Community
Number analyzed (Participants) | 1480 | 1471 | 0
Number analyzed (communities) | 9 | 9 | 0
number of minutes per day within bouts o | -1.35 (1.82) | -0.18 (1.80) |
Statistical Analysis 1: Comparison: CHL Program vs Control Community; Intervention vs control comparing 24 months to baseline; Test type: Superiority — Hierarchical linear model accounting for randomization of communities and clustering of children within communities in strata of jurisdictions weighted for number of children less than age 10 in communities. Chi-square test accounts for degrees of freedom based on number of communities; p = 0.68, Regression, Linear; Mean Difference (Final Values) = -1.17

8. Secondary Outcome: Change in Sedentary and Light Physical Activity
Description: number of minutes per day within bouts of 5 minutes averaged over 4 to 6 days of accelerometer usage
Time Frame: Baseline, 24 months
Population: Children 2 to 8 randomized to CHL program or Control Community. Temporal community not assessed for physical activity.
Measure: Mean (Standard Error); unit: number of minutes per day within bouts o
Units Other Than Participants: communities
Arm/Group | CHL Program | Control Community | Temporal Community
Number analyzed (Participants) | 1480 | 1471 | 0
Number analyzed (communities) | 9 | 9 | 0
number of minutes per day within bouts o | 1.78 (3.96) | -1.64 (3.90) |
Statistical Analysis 1: Comparison: CHL Program vs Control Community; Intervention vs control comparing 24 months to baseline; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.55, Regression, Linear; Mean Difference (Final Values) = 3.42

9. Secondary Outcome: Change in Screen Time
Description: Hours per day spent in screen activity
Time Frame: Change from Baseline to 24 months
Population: Children 2 to 8 randomized to CHL program or Control Community. Temporal community not assessed for screen time.The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.
Measure: Mean (Standard Error); unit: hours per day
Units Other Than Participants: communities
Groups:
- Temporal Community: Communities assessed for temporal change in anthropometry.
Arm/Group | CHL Program | Control Community | Temporal Community
Number analyzed (Participants) | 2859 | 2786 | 0
Number analyzed (communities) | 9 | 9 | 0
hours per day | -0.2 (0.18) | 0.3 (0.22) |
Statistical Analysis 1: Comparison: CHL Program vs Control Community; Intervention vs control comparing 24 months to baseline; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.11, Regression, Linear; Mean Difference (Final Values) = -0.5

10. Secondary Outcome: Sleep Disturbance Score
Description: Tayside sleep scale; minimum is 1, maximum is 9, where higher is worse. lower score is less disturbance (range is 1-9) Tayside Children's Sleep Questionnaire by McGreavey JA, Donnan PT, Pagliari HC, Sullivan FM.The Tayside children's sleep questionnaire: a simple tool to evaluate sleep problems in young children. Child Care Health Dev. 2005 Sep;31(5):539-44.
Time Frame: Change from Baseline to 24 months
Population: Children 2 to 8y randomized to CHL program or Control Community. Temporal community not assessed for sleep disturbance.The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: communities
Arm/Group | CHL Program | Control Community | Temporal Community
Number analyzed (Participants) | 2859 | 2786 | 0
Number analyzed (communities) | 9 | 9 | 0
units on a scale | -0.4 (0.35) | 0.3 (0.19) |
Statistical Analysis 1: Comparison: CHL Program vs Control Community; mixed model adjusting for age and sex and cluster of community and strata of jurisdiction; intervention vs control comparing 24 months to baseline; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.08, Regression, Linear; Mean Difference (Final Values) = -0.7

11. Secondary Outcome: Change in Water Intake
Description: cups per day, determined from 2 random days of food records and weighted for weekend and weekday. The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.
Time Frame: Change from Baseline to 24 months
Population: Children 2 to 8 randomized to CHL program or Control Community. Temporal community not assessed for water intake.
Measure: Mean (Standard Error); unit: cups per day
Units Other Than Participants: communities
Arm/Group | CHL Program | Control Community | Temporal Community
Number analyzed (Participants) | 2859 | 2786 | 0
Number analyzed (communities) | 9 | 9 | 0
cups per day | 0.07 (0.06) | 0.11 (0.04) |
Statistical Analysis 1: Comparison: CHL Program vs Control Community; Intervention vs control comparing 24 months to baseline; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.71, Regression, Linear; Hierarchical model; Mean Difference (Final Values) = -0.04

12. Secondary Outcome: Change in Fruit Intake
Description: cups per day, determined from 2 random days of food records and weighted for weekend and weekday
Time Frame: Change from baseline to 24 months
Population: Children 2 to 8 randomized to CHL program or Control Community. Temporal community not assessed for fruit intake.
Measure: Mean (Standard Error); unit: cups per day
Units Other Than Participants: communities
Arm/Group | CHL Program | Control Community | Temporal Community
Number analyzed (Participants) | 2859 | 2786 | 0
Number analyzed (communities) | 9 | 9 | 0
cups per day | -0.07 (0.03) | -0.05 (0.02) |
Statistical Analysis 1: Comparison: CHL Program vs Control Community; Intervention vs control comparing 24 months to baseline; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.54, Regression, Linear; Hierarchical model; Mean Difference (Final Values) = -0.02

13. Secondary Outcome: Change in Vegetable Intake
Description: cups per day, determined from 2 random days of food records and weighted for weekend and weekday
Time Frame: Change from baseline to 24 months
Population: Children 2 to 8y randomized to CHL program or Control Community. Temporal community not assessed for vegetable intake.
Measure: Mean (Standard Error); unit: cups per day
Units Other Than Participants: communities
Arm/Group | CHL Program | Control Community | Temporal Community
Number analyzed (Participants) | 2859 | 2786 | 0
Number analyzed (communities) | 9 | 9 | 0
cups per day | -0.01 (0.02) | 0 (0.01) |
Statistical Analysis 1: Comparison: CHL Program vs Control Community; Intervention vs control comparing 24 months to baseline; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.90, Regression, Linear; Mean Difference (Final Values) = -0.01

14. Secondary Outcome: Change in Metabolic Equivalents (METs) Per Day
Description: number of minutes per day within bouts of 5 minutes averaged over 4 to 6 days of accelerometer usage
Time Frame: Baseline, 24 months
Population: Children 2 to 8y randomized to CHL program or Control Community. Temporal community not assessed for accelerometry.
Measure: Mean (Standard Error); unit: number of minutes per day within bouts o
Units Other Than Participants: communities
Groups:
- Temporal Community: Communities assessed for temporal changes in anthropometry.
Arm/Group | CHL Program | Control Community | Temporal Community
Number analyzed (Participants) | 1480 | 1471 | 0
Number analyzed (communities) | 9 | 9 | 0
number of minutes per day within bouts o | -0.29 (0.09) | -0.24 (0.09) |
Statistical Analysis 1: Comparison: CHL Program vs Control Community; Intervention vs control comparing 24 months to baseline; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.71, Regression, Linear; Mean Difference (Final Values) = -0.05

15. Secondary Outcome: Change in Hours of Sleep Per Day
Description: Sleep hours per day measure by questionnaire as reported by caregiver.
Time Frame: change from baseline to 24 months
Population: Children 2-8y in the selected Pacific communities.
Measure: Mean (Standard Error); unit: hours per day
Units Other Than Participants: communities
Arm/Group | CHL Program | Control Community | Temporal
Number analyzed (Participants) | 2859 | 2786 | 2726
Number analyzed (communities) | 9 | 9 | 9
hours per day | 0.07 (0.16) | 0.25 (0.17) | 0.09 (0.17)
Statistical Analysis 1: Comparison: CHL Program vs Control Community vs Temporal; Intervention vs control comparing 24 months to baseline; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.48, Regression, Linear — intervention vs control communities; Mean Difference (Final Values) = -0.18

16. Primary Outcome: Prevalence of Acanthosis Nigricans
Description: as for outcome 3
Time Frame: Baseline, 78 months
Population: as for outcome 3
Measure: Mean (Standard Error); unit: percentage of 2-8 yo children
Units Other Than Participants: communities
Arm/Group | CHL Program | Control Community | Temporal Community
Number analyzed (Participants) | 2017 | 1970 | 0
Number analyzed (communities) | 9 | 9 | 0
percentage of 2-8 yo children | -4.1 (0.79) | -0.5 (0.96) |
Statistical Analysis 1: Comparison: CHL Program vs Control Community; intervention vs control. The children from each community recruited each time were NOT the same children. The number of communities is consistent across time; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.01, Regression, Logistic — [p-value comment as in outcome 1, analysis 2]; Hierarchical model; differences in prevalence = -3.6

17. Secondary Outcome: Change in Sugar Sweetened Beverage Intake
Description: cups per day, determined from 2 random days of food records and weighted for weekend and weekday
Time Frame: change from baseline to 78 months
Population: as for outcome 6
Measure: Mean (Standard Error); unit: cups per day
Units Other Than Participants: communities
Arm/Group | CHL Program | Control Community | Temporal Community
Number analyzed (Participants) | 2017 | 1970 | 0
Number analyzed (communities) | 9 | 9 | 0
cups per day | -0.05 (0.07) | -0.14 (0.08) |
Statistical Analysis 1: Comparison: CHL Program vs Control Community; [analysis description as in outcome 16, analysis 1]; Test type: Superiority — Hierarchical; p = 0.44, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = 0.09

18. Secondary Outcome: Change in Screen Time
Description: Hours per day spent in screen activity
Time Frame: change from Baseline to 78 months
Population: as for outcome 9
Measure: Mean (Standard Error); unit: hours per day
Units Other Than Participants: communities
Arm/Group | CHL Program | Control Community | Temporal Community
Number analyzed (Participants) | 2017 | 1970 | 0
Number analyzed (communities) | 9 | 9 | 0
hours per day | 0.006 (0.01) | 0.10 (0.02) |
Statistical Analysis 1: Comparison: CHL Program vs Control Community; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.81, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = 0.16

19. Secondary Outcome: Sleep Disturbance Score
Description: as for outcome 10
Time Frame: Change from baseline to 78 months, The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.
Population: Children 2 to 8y randomized to CHL program or Control Community. Temporal community not assessed for sleep disturbance.
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: communities
Arm/Group | CHL Program | Control Community | Temporal Community
Number analyzed (Participants) | 2017 | 1970 | 0
Number analyzed (communities) | 9 | 9 | 0
units on a scale | 1.83 (0.02) | 1.46 (0.05) |
Statistical Analysis 1: Comparison: CHL Program vs Control Community; [analysis description as in outcome 1, analysis 2]; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.68, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = 0.37 — [estimate comment as in outcome 4, analysis 1]

20. Secondary Outcome: Change in Water Intake
Description: cups per day, determined from 2 random days of food records and weighted for weekend and weekday
Time Frame: change from baseline to 78 months.The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.
Population: Children 2 to 8 randomized to CHL program or Control Community. Temporal community not assessed for water intake.The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.
Measure: Mean (Standard Error); unit: cups per day
Units Other Than Participants: communities
Arm/Group | CHL Program | Control Community | Temporal Community
Number analyzed (Participants) | 2017 | 1970 | 0
Number analyzed (communities) | 9 | 9 | 0
cups per day | 0.02 (0.03) | 0 (0.02) |
Statistical Analysis 1: Comparison: CHL Program vs Control Community; [analysis description as in outcome 16, analysis 1]; Test type: Superiority — Hierarchical model. The children from each community recruited each time were NOT the same children. The number of communities is consistent across time; p = 0.69, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = 0.02

21. Secondary Outcome: Change in Fruit Intake
Description: cups per day, determined from 2 random days of food records and weighted for weekend and weekday
Time Frame: change from baseline to 78 months
Population: Children 2 to 8 randomized to CHL program or Control Community. Temporal community not assessed for fruit intake.
Measure: Mean (Standard Error); unit: cups per day
Units Other Than Participants: communities
Arm/Group | CHL Program | Control Community | Temporal Community
Number analyzed (Participants) | 2017 | 1970 | 0
Number analyzed (communities) | 9 | 9 | 0
cups per day | 0.02 (0.06) | -0.19 (0.10) |
Statistical Analysis 1: Comparison: CHL Program vs Control Community; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — [test comment as in outcome 20, analysis 1]; p = 0.11, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Final Values) = 0.21 — [estimate comment as in outcome 4, analysis 1]

22. Secondary Outcome: Change in Vegetable Intake
Description: cups per day, determined from 2 random days of food records and weighted for weekend and weekday
Time Frame: change from baseline to 78 months
Population: Children 2 to 8y randomized to CHL program or Control Community. Temporal community not assessed for vegetable intake.
Measure: Mean (Standard Error); unit: cups per day
Units Other Than Participants: communities
Arm/Group | CHL Program | Control Community | Temporal Community
Number analyzed (Participants) | 2017 | 1970 | 0
Number analyzed (communities) | 9 | 9 | 0
cups per day | 0 (0.05) | -0.06 (0.04) |
Statistical Analysis 1: Comparison: CHL Program vs Control Community; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — [test comment as in outcome 20, analysis 1]; p = 0.40, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Final Values) = 0.06

23. Secondary Outcome: Change in Hours of Sleep Per Day
Description: Sleep hours per day measure by questionnaire as reported by caregiver.
Time Frame: change from baseline to 78 months
Population: Children 2-8y in the selected Pacific communities.The children from each community recruited each time were NOT the same children. The number of communities is consistent across time.
Measure: Mean (Standard Error); unit: hours per day
Units Other Than Participants: communities
Arm/Group | CHL Program | Control Community | Temporal
Number analyzed (Participants) | 2017 | 1970 | 1811
Number analyzed (communities) | 9 | 9 | 9
hours per day | 0.2 (0.18) | 0 (0.11) | 0.01 (0.2)
Statistical Analysis 1: Comparison: CHL Program vs Control Community; [analysis description as in outcome 16, analysis 1]; Test type: Superiority — [test comment as in outcome 20, analysis 1]; p = 0.37, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = 0.20
Statistical Analysis 2: Comparison: CHL Program vs Temporal; Intervention vs temporal.The children from each community recruited each time were NOT the same children. The number of communities is consistent across time; Test type: Superiority — Hierarchical model.The children from each community recruited each time were NOT the same children. The number of communities is consistent across time; p = 0.51, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = 0.18

ADVERSE EVENTS:
Time Frame: The children representing the communities were observed for the assessment periods only.
Groups:
- Delayed Optimized CHL Program: Control community that participated in community engagement process and received delayed optimized program.
Arm/Group | CHL Program | Delayed Optimized CHL Program | Temporal
All-Cause Mortality (participants affected / at risk) | 0/3359 | 0/3265 | 0/3216
Serious Adverse Events (participants affected / at risk) | 0/3359 | 0/3265 | 0/3216
Other Adverse Events (participants affected / at risk) | 0/3359 | 0/3265 | 0/3216

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No